CLINICAL TRIAL: NCT00313287
Title: A Double-Blind, Randomized, Parallel, Placebo-Controlled Phase III Study to Evaluate the Safety and Antiviral Activity of Clevudine 30 mg QD in Patients Chronically Infected With Hepatitis B Virus
Brief Title: Safety and Antiviral Activity Study of Clevudine 30 mg QD in Patient With Chronic HBV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-FMAU-301
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2006-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: clevudine

SUMMARY:
The purpose of this study is to determine safety and efficacy of 30 mg daily dose of clevudine (L-FMAU) at 24 weeks of treatment in patients with chronic HBV.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were between 18 and 60, inclusive.
2. Patients with HBV DNA ³1 x 106 copies/mL within 30 days of baseline.
3. Patients who were documented to be HBsAg positive for > 6 months. (The documentation of positive HBsAg for the previous 6 months included previous laboratory reports of HBsAg positive or HBeAg positive at least 6 month ago or IgM anti-HBc negative and IgG anti-HBc positive at screening).
4. Patients who were HBeAg positive.
5. Patients with ALT levels which were in the range of ≥1.2 and < 15 times of the upper limit of normal (x ULN) and bilirubin levels less than 2.0 mg/dL, prothrombin time of less than 1.7 (INR), and a serum albumin level of at least 3.5 g/dL.
6. Women of child bearing potential with a negative serum (β-HCG) pregnancy test taken within 14 days of starting therapy.
7. Patients who were able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patients who were currently receiving antiviral, immunomodulatory or corticosteroid therapy.
2. Patients previously treated with lamivudine, lobucavir, famciclovir, adefovir or any other investigational nucleoside for HBV infection.
3. Previous treatment with interferon that had ended less than 6 months prior to the screening visit.
4. Patients with a history of ascites, variceal hemorrhage or hepatic encephalopathy.
5. Patients co-infected with HCV, HDV or HIV.
6. Patients with clinical evidence of liver mass or with alpha-fetoprotein > 50 ng/mL
7. Patients who were pregnant or breast-feeding.
8. Patients who were unwilling to use an "effective" method of contraception during the treatment and for up to 3 months after cessation of therapy. For males, condoms should be used. Females had to be surgically sterile (via hysterectomy or bilateral tubal ligation) or post-menopausal or using at least medically acceptable barrier method of contraception ( i.e. IUD, barrier methods with spermicide or abstinence)
9. Patients with a clinically relevant history of abuse of alcohol or drugs.
10. Patients with a significant gastrointestinal, renal, hepatic (decompensated), bronchopulmonary, biliary diseases except asymptomatic GB stone, neurological, cardiovascular, oncologic or allergic disease.

    The patients with a benign tumor were excluded if judged by an investigator that the continuation of study would be interfered by benign tumor.
11. Patients with creatinine clearance less than 60mL/min as estimated by the following formula :

(140-age in years) (body weight [kg]) (72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Patients who were found to have YMDD HBV DNA polymerase mutation at baseline were to be excluded from the overall efficacy evaluation and analyzed separately. They were to be included in the overall safety evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180
Dates: Start 2003-06; Study Completion 2004-11

PRIMARY OUTCOMES:
Efficacy:change from baseline in HBV DNA (log10) at Week 24
Safety: clinically measured adverse events, abnormality of laboratory tests and abnormality of vital signs.

SECONDARY OUTCOMES:
Efficacy:
Proportion of patients with HBV DNA below the assay Limit of Detection
Proportion of patients with HBeAg loss and/or seroconversion (HBeAg loss and HBeAb gain)
Proportion of ALT normalization

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Suk Lee, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (33):
- South Korea (33):
  - St. Mercy's Hospital, Bupyoung-dong, Bupyoung-gu, Incheon
  - Pusan Paik Hospital, Gaegeum-dong, Busan
  - Kangbuk Samsung Hospital, Pyoung-dong, Chongro-gu, Seoul
  - Keimyumg University Dongsan Medical Center, Jung-gu, Daegu
  - Kyungpook National University Medical Hospital, Jung-gu, Daegu
  - Chonnam National University Hospital, Hak-1-dong, Dong-gu, Gwangju-si
  - Korea University Guro Hospital, Seoul, Gro-gu
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungnam National University Hospital, Daesadong, Jung-gu, Daechon
  - Inha University Hospital, Sinhŭng-dong, Jung-gu, Incheon
  - Seoul Asan Medical Center, Pungnap-dong, Kangnam-gu, Seoul
  - Yongdong Severance Hospital, Togok-tong, Kangnam-gu, Seoul
  - National Cancer Center, Ilsan-gu, Kyounggi-do
  - St. Holly Family Mary's Hospital, Pucheon, Kyounggi-do
  - Pochon CHA University Hospital, Seongnam-gu, Kyounggi-do
  - Yeungnam University Medical Center, Dae Myoung-dong, Nam-gu, Taegu
  - Korea Cancer Center Hospital, Gongneungdong, Nowon-gu, Seoul
  - Nowon Eulji Hospital, Hagyeil-tong, Nowon-gu, Seoul
  - St. Vincent's Hospital, Chi-dong, Paldal-gu, Suwon
  - Pusan National University Hospital, Ami-dong, Seo-gu, Pusan
  - Kosin Medical Center, Amnam-dong, Seo-gu, Pusan
  - KangNam St. Mary's Hospital, Banpo-dong, Seocho-gu, Seoul
  - Severance Hospital, Shinchon- Dong, Seodaemun-gu, Seoul
  - Seoul Paik Hospital, Jeo-dong, Seoul
  - Samsung Medical Center, Ilwon-dong, Songpa-gu, Seoul
  - Korea University Anam Hospital, Anam-dong, Sungbuk-ku, Seoul
  - Ehwa Womans University Mokdong Hospital, Mokdong, Yangcheon-gu, Seoul
  - Kangnam Sacred Heart Hospital, Daelim-dong, Yongdeungpo-gu, Seoul
  - Soon Chun Hyang University Hospital, Hannam-dong, Yongsan-gu, Seoul
  - St. Mary's Hospital, Seoul, Yungdungpo-Gu
  - Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul